CLINICAL TRIAL: NCT05464459
Title: A Prospective Case Series to Evaluate the Outcomes and Acceptability of a Novel Surgical Technique of Pyrocarbon Interposition Arthroplasty of the Elbow, in Young Patients With Severe Arthritis.
Brief Title: Pyrocarbon Interposition Arthroplasty of the Elbow
Acronym: HAPY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wrightington, Wigan and Leigh NHS Foundation Trust (Other)
Collaborators: Edge Hill University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAPY
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis of Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HAPY interposition elbow replacement (Experimental): HAPY is a pyrocarbon sphere for use as an interposition joint replacement. In this study, the implant is being used as a novel procedure in the Elbow (outside approved label usage)
  Interventions: Procedure: Novel elbow procedure

INTERVENTIONS:
Procedure: Novel elbow procedure — A general anaesthetic plus upper limb nerve block is used with no tourniquet. Antibiotics and tranexamic acid are administered intravenously prior to procedure. Skin prepared by standard technique with alcoholic chlorhexidine. A posterior midline incision is made and lateral paraolecranon approach made to the elbow joint. Lateral ligament complex released for access and repaired at the end of the procedure. A 5mm high speed burr and HAPY burr instrument prepares the distal humerus. The trochlea spool and/or capitellum are resected to receive Pyrocarbon spherical prosthesis, size determined from pre-operative planning. The greater sigmoid notch is prepared in a similar manner with burr. A trial prosthesis is used to assess joint movement/stability before the Pyrocarbon spherical spacer inserted. Wound closed in layers with heavy vicryl. Skin closure with subcutaneous monocryl. Physiotherapist advice within 24 hours and immediate active mobilisation is commenced as comfort allows.

SUMMARY:
The current study will be a prospective observational study (or collective case study in a small, carefully selected cohort of consenting patients with advanced arthritis. This study would be classified as a stage I study according the IDEAL framework for surgical innovation

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the elbow is associated with pain and loss of motion, which can have a dramatic impact on overall upper limb function due to the inability to position the hand to carry out activities of daily living. OA is characterised by osteophyte formation of the olecranon, coronoid and olecranon fossae, whilst the ulnohumeral and radiohumeral joint spaces may be relatively well preserved. The osteophytes cause terminal extension and flexion pain and impingement, whilst the limited arc of movement is often relatively pain-free. Loose bodies are also commonly present and can cause mechanical locking. Pain throughout the limited range of movement however, indicates joint destruction. This can be confirmed radiographically, which in contrast to the typical OA presentation described above, shows articular cartilage loss with narrowing or obliteration of the entire joint space, not usually seen in primary osteoarthritis. The pathologies in which loss of joint space is more commonly seen are post-septic arthritis, post-traumatic arthritis and inflammatory arthritis.

Total elbow arthroplasty (TEA) is thought to be an effective treatment for a range of pathologies including rheumatoid arthritis, late stage primary osteoarthritis, acute fracture and post-traumatic arthritis. However, it has been reported in the literature that younger patients undergoing TEA may experience earlier failure of the implant and higher complication rates. This is thought to be linked to higher functional demands placed on the implant due to greater occupational loading or participation in more demanding leisure activities. For this reason, other viable alternative to TEA are being sought by surgeons for younger patients with high functional demands.

Interposition arthroplasty has been proposed as an alternative to TEA for younger patients in the literature with various surgical techniques described. According to Thomas, the basic principle of interposition arthroplasty of the elbow is to perform a resection of the opposing bone ends and place something in between the distal humerus and the olecranon, which will then theoretically allow movement to occur without painful grinding of the joint.

Two of the major risks of TEA are aseptic loosening and periprosthetic infection. In the event of a significant joint infection, revision of the TEA procedure is often necessary and may be performed as a two-stage operation. Initially the prosthesis is removed and the infection is treated, a process that often involves the use of an antibiotic-impregnated spacer and oral antibiotics. If appropriate, once the infection is eradicated, a new prosthesis will be implanted. Cases have however been documented in the literature where the patients in receipt of spherical antibiotic cement spacers are satisfied with the movement and pain relief provided by the spacer, and subsequently decline re-implantation of a second prosthesis and. This has led the current author to question whether interposition arthroplasty using a spherical joint spacer may be a viable alternative to TEA in young patients with higher functional demands in whom there is a greater risk of premature aseptic loosening after TEA.

Pyrocarbon interposition implants have been successfully used in the small joints of the hand, wrist and foot, and more recently their use has been trialed in the shoulder with acceptable outcomes . Pyrocarbon is deemed an ideal material for the manufacture of orthopaedic implants due to its strength, resistance to wear and resistance to fatigue. It is also stated in the literature that there have been no reports of periarticular infiltration or reaction to pyrocarbon particles transmitted by the blood or lymphatic systems into organs such as the brain, kidneys or liver.

In the current study, we propose to perform interposition arthroplasty of the elbow using a spherical pyrocarbon implant normally used in the hand and wrist ('HAPY' pyrocarbon sphere, Wright Medical, USA), in a small case series of specially selected young patients with advanced arthritis who would otherwise require a total elbow arthroplasty.

Eligible patients attending the current author's clinic with advanced arthritis of the elbow, who are unsuitable for TEA due to their young age and high functional demands, will be invited to be part of the study. They will undergo the same pre and post-operative radiographic investigations as those undergoing TEA; A/P and lateral X-Ray views of the elbow at approximately 3 weeks, 3 months, 6 months, 12 months and 24 months. They will also complete patient reported outcome measures (PROMs) both pre-operatively, and at each of their post-operative clinic visits, as per routine practice within the host NHS Trust. Each of the PROMs to be used in this study will be a validated measure of upper limb function suitable for use in those with elbow pathology. An 11 point numerical rating scale for measurement of pain level will also be completed at each time-point in addition to goniometric measurement of elbow range of movement using a standardised technique and recording of adverse events. It is usual practice within the host NHS Trust for patients undergoing TEA to be reviewed following surgery at approximately 3 weeks, 3 months, 6 months, one year and 2 years. The same approximate follow-up schedule will be followed for patients undergoing the study procedure unless early problems are identified and there is a clinical need for more frequent follow-up assessment.

The protocol has been sent for external independent scientific review. The outcome of which has been enclosed alongside this protocol for review by the committee.

It will be made clear to all participants that pyrocarbon interposition arthroplasty of the elbow is an innovative and novel procedure and that the alternatives to this treatment would be TEA or continued conservative management. If the procedure fails to provide an acceptable outcome, the patient would then be offered a revision to a TEA. The previous interposition arthroplasty should not compromise a subsequent total elbow replacement as the bone resection is limited.

The previous literature relating to the use of spherical cement spacers in the elbow and the use of pyrocarbon interposition arthroplasty in other joints, leads us to believe that the proposed procedure in this study would prove a viable alternative for young patients with advanced arthritis of the elbow joint. However, for patient safety, a data monitoring committee will scrutinise the early data and if the complication rate is unacceptable or outcome unsatisfactory, the study will be terminated. The findings of this study, regardless of the number of participants or the success of the procedure, will be submitted for publication to further advance this field of orthopaedic practice.

The study data will be subject to internal scrutiny at 6 monthly intervals by colleagues within the upper limb unit at Wrightington, and external scrutiny by an external expert in the field.

ELIGIBILITY:
Inclusion Criteria:

* Medically fit for surgery
* Advanced osteoarthritis, post-traumatic arthritis, or post-septic arthritis
* Severe inflammatory arthritis without severe bone destruction - Larsen grade III or less
* Failed conservative treatment
* Unsuitable for TEA due to high functional demands

Exclusion Criteria:

* Severe inflammatory arthritis with severe bone destruction
* Arthritis suitable for treatment with arthroscopic debridement.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and acceptability | 24 months
  The principal research objective is to assess the safety and acceptability of interposition arthroplasty of the elbow using a spherical pyrocarbon implant in a prospective consecutive case series of carefully selected patients.

SECONDARY OUTCOMES:
Motion Analysis | 24 months
  Secondary Objective using motion analysis (special equipment to measure small movements and changes in elbow biomechanics) will be to quantify elbow joint Range of Movement and stability pre-operatively, and at 3- and 6-months post-operatively following interposition elbow arthroplasty and to compare this to a sex-matched group of patients after total elbow replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Watts, Principal Investigator — Wrightington, Wigan & Leigh Teaching Hospitals NHS Foundation Trust
Locations (1):
- Wrightington, Wigan & Leigh Teaching Hospitals NHS Foundation Trust, Wigan, United Kingdom

IPD SHARING:
Plan to Share IPD: No